CLINICAL TRIAL: NCT00703170
Title: Phase I Study of Pegylated Liposomal Doxorubicin and Temsirolimus in Resistant Solid Malignancies
Brief Title: Phase I Study of DOXIL and Temsirolimus in Resistant Solid Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-0447
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Last update posted 2013-05-24 (Estimated); Status verified 2013-05

CONDITIONS: Resistant Solid Malignancies
MeSH Terms: interventions — temsirolimus; liposomal doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dose Level 1 (original) (Experimental): Temsirolimus IV 20 mg weekly
  Pegylated liposomal doxorubicin IV 30 mg/m2 once every 4 weeks
  Interventions: Drug: Temsirolimus; Drug: Pegylated liposomal doxorubicin
- Dose Level 1 (revised) (Experimental): Temsirolimus IV 20 mg weekly
  Pegylated liposomal doxorubicin IV 25 mg/m2 once every 4 weeks
  Interventions: Drug: Temsirolimus; Drug: Pegylated liposomal doxorubicin
- Dose Level 2 (Experimental): Temsirolimus IV 25 mg weekly
  Pegylated liposomal doxorubicin IV 25 mg/m2 once every 4 weeks
  Interventions: Drug: Temsirolimus; Drug: Pegylated liposomal doxorubicin

INTERVENTIONS:
Drug: Temsirolimus
  Other Names: Torisel; CCI-779
Drug: Pegylated liposomal doxorubicin
  Other Names: DOXIL

SUMMARY:
Rationale:

The Mammalian Target of Rapamycin (mTOR) is a large polypeptide serine/threonine kinase of 289 kDa; kinases have been shown to be important regulators of cancer cell cycle, proliferation, invasion, and angiogenesis, and mTOR has been shown to have a key role in the signaling of malignant cell growth, proliferation, differentiation, migration, and survival. Inhibition of mTOR would result in arrest of cell growth in the G1 phase of the cell cycle.

Temsirolimus (CCI-779) is a soluble ester analogue of rapamycin (sirolimus) which has shown impressive in vitro and in vivo cytostatic activity in selectively inhibiting mTOR. In animal models, temsirolimus has demonstrated an impressive cytostatic effect on a wide variety of cancer cells. In vitro, it inhibited the growth of human T-cell leukemia, glioblastoma, melanoma, prostate, breast, renal cell, and pancreatic cells, all of which showed particular sensitivity to temsirolimus, with significant growth inhibition at concentrations of less that 0.01micrometer. In Phase I trials, temsirolimus has been investigated as a single agent on a weekly schedule as well as daily for 5 days every other week, and evidence of activity was observed over the entire dose range (15 - 220 mg/m2) in patients with both breast and renal cancer. There was no apparent relationship between exposure and clinical benefit, suggesting that the inhibition of mTOR may be achieved at doses well below dose levels that result in dose limiting toxicities. Major tumor responses were noted in Phase I trials in patients previously treated with lung, breast, renal as well as neuroendocrine tumors. Minor responses were noted in soft tissue sarcoma, endometrial, and cervical carcinoma.

Pegylated liposomal doxorubicin has been FDA approved for use in refractory metastatic ovarian cancer and AIDS-related Kaposi's Sarcoma. It has also been shown to be effective in previously treated metastatic breast cancer.

Combination studies in preclinical models suggest that rapamycin and its analogues are at least additive in effect with standard chemotherapy and radiation. In addition, studies in breast cancer cell lines suggest that the mTOR inhibitors may reverse resistance to anti-estrogen agents. Thus, we are proposing that the combination of temsirolimus and liposomal doxorubicin will be highly effective in metastatic solid tumor malignancies.

Objectives:

Primary

* To define the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of temsirolimus in combination with pegylated liposomal doxorubicin in patients with resistant solid malignancies.
* To determine the incidence and severity of other toxicities of temsirolimus in combination with pegylated liposomal doxorubicin in patients with resistant solid malignancies.

Secondary

* To assess the pharmacokinetic profile of temsirolimus in combination with pegylated liposomal doxorubicin.
* To determine any anti-tumor activity and response to the combination of temsirolimus and pegylated liposomal doxorubicin in treatment of patients with resistant solid malignancies.

ELIGIBILITY:
Inclusion and Exclusion Criteria:

* Patients must have a histologically or cytologically proven solid malignancy which is resistant to conventional therapy or for which no effective therapy is known.
* Patients with measurable or non-measurable disease are eligible for entry to this study. In addition, patients without measurable or non-measurable disease are also eligible.
* Patients must have recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study. No chemotherapy or radiotherapy may be given within 4 weeks prior to the start of protocol treatment.
* Patients must be ≥18 years old.
* ECOG 0-2 at study entry.
* Patients must have a life expectancy of greater than 8 weeks.
* Required Laboratory Values:
* absolute neutrophil count ≥1,500/mm3
* platelets ≥100,000/mm3
* hemoglobin ≥9.0 g/dL
* total bilirubin ≤1.5 x ULN
* AST(SGOT)/ALT(SGPT) ≤1.5 x ULN (≤2.5 x ULN for patients with liver metastases)
* alkaline phosphatase ≤2.5 x ULN
* creatinine ≤1.5 x ULN OR
* creatinine clearance ≥60 mL/min/1.732 for patients with creatinine levels above 2.0 mg/dl
* serum cholesterol ≤350 mg/dL /9.0 mmol/L (fasting)
* triglycerides ≤400 mg/dL (fasting)*
* albumin ≥3.0 mg/dL
* PT/INR ≤1.5, unless the patient is on full dose warfarin or stable dose of LMW heparin with a therapeutic INR of >1.5 - ≤3 *Patients with triglyceride levels >400 mg/dL can be started on lipid lowering agents and reevaluated within 1 week. If levels go to ≤400 mg/dL, they can be considered for the trial and continue the lipid lowering agents.
* Temsirolimus is primarily metabolized by CYP3A4. Patients cannot be receiving enzyme-inducing antiepileptic drugs (EIAEDs; e.g., phenytoin, carbamazepine, phenobarbital) nor any other CYP3A4 inducer such as rifampin or St. John's wort, as these may decrease temsirolimus levels.
* Patients with known hypersensitivity reactions to macrolide antibiotics (such as erythromycin, clarithromycin, and azithromycin) are not eligible for this trial.
* Patients must have a normal left ventricular ejection fraction (LVEF ≥50%) by MUGA scan.
* For all sexually active patients, the use of adequate contraception (hormonal or barrier method of birth control) will be required prior to study entry and for the duration of study participation. Non-pregnant status will be determined in all women of childbearing potential. Pregnant and nursing women are not eligible.
* Patients receiving anti-retroviral therapy (HAART) for HIV infection are excluded from the study because of possible pharmacokinetic interactions.
* Patients must not have active CNS disease.
* Patients must have recovered from uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris or cardiac arrhythmia.
* Patients must have signed a Washington University, Human Research Protection Office (HRPO) approved informed consent. The patient should not have any serious medical or psychiatric illness that would prevent either the giving of informed consent or the receipt of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-03; Primary Completion 2011-06 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
To define the maximum tolerated dose (MTD) and dose-limiting toxicities (DLT) of temsirolimus in combination with pegylated liposomal doxorubicin in patients with resistant solid malignancies. | After completion of cycle 1 by all patients
To determine the incidence and severity of other toxicities of temsirolimus in combination with pegylated liposomal doxorubicin in patients with resistant solid malignancies. | 30 days after completion of treatment

SECONDARY OUTCOMES:
To assess the pharmacokinetic profile of temsirolimus in combination with pegylated liposomal doxorubicin. | 2 years
To determine any anti-tumor activity and response to the combination of temsirolimus and pegylated liposomal doxorubicin in treatment of patients with resistant solid malignancies. | Completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Joel Picus, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Background] Vignot S, Faivre S, Aguirre D, Raymond E. mTOR-targeted therapy of cancer with rapamycin derivatives. Ann Oncol. 2005 Apr;16(4):525-37. doi: 10.1093/annonc/mdi113. Epub 2005 Feb 22. PMID 15728109
- [Background] Sabers CJ, Martin MM, Brunn GJ, Williams JM, Dumont FJ, Wiederrecht G, Abraham RT. Isolation of a protein target of the FKBP12-rapamycin complex in mammalian cells. J Biol Chem. 1995 Jan 13;270(2):815-22. doi: 10.1074/jbc.270.2.815. PMID 7822316
- [Background] Lorenz MC, Heitman J. TOR mutations confer rapamycin resistance by preventing interaction with FKBP12-rapamycin. J Biol Chem. 1995 Nov 17;270(46):27531-7. doi: 10.1074/jbc.270.46.27531. PMID 7499212
- [Background] Janus A, Robak T, Smolewski P. The mammalian target of the rapamycin (mTOR) kinase pathway: its role in tumourigenesis and targeted antitumour therapy. Cell Mol Biol Lett. 2005;10(3):479-98. PMID 16217558
- [Background] O'Reilly KE, Rojo F, She QB, Solit D, Mills GB, Smith D, Lane H, Hofmann F, Hicklin DJ, Ludwig DL, Baselga J, Rosen N. mTOR inhibition induces upstream receptor tyrosine kinase signaling and activates Akt. Cancer Res. 2006 Feb 1;66(3):1500-8. doi: 10.1158/0008-5472.CAN-05-2925. PMID 16452206
- [Background] Oldham S, Hafen E. Insulin/IGF and target of rapamycin signaling: a TOR de force in growth control. Trends Cell Biol. 2003 Feb;13(2):79-85. doi: 10.1016/s0962-8924(02)00042-9. PMID 12559758
- [Background] Bianco R, Melisi D, Ciardiello F, Tortora G. Key cancer cell signal transduction pathways as therapeutic targets. Eur J Cancer. 2006 Feb;42(3):290-4. doi: 10.1016/j.ejca.2005.07.034. Epub 2006 Jan 11. PMID 16376541
- [Background] Sansal I, Sellers WR. The biology and clinical relevance of the PTEN tumor suppressor pathway. J Clin Oncol. 2004 Jul 15;22(14):2954-63. doi: 10.1200/JCO.2004.02.141. PMID 15254063
- [Background] DeGraffenried LA, Fulcher L, Friedrichs WE, Grunwald V, Ray RB, Hidalgo M. Reduced PTEN expression in breast cancer cells confers susceptibility to inhibitors of the PI3 kinase/Akt pathway. Ann Oncol. 2004 Oct;15(10):1510-6. doi: 10.1093/annonc/mdh388. PMID 15367412
- [Background] Manning BD, Tee AR, Logsdon MN, Blenis J, Cantley LC. Identification of the tuberous sclerosis complex-2 tumor suppressor gene product tuberin as a target of the phosphoinositide 3-kinase/akt pathway. Mol Cell. 2002 Jul;10(1):151-62. doi: 10.1016/s1097-2765(02)00568-3. PMID 12150915
- [Background] Hidalgo M, Rowinsky EK. The rapamycin-sensitive signal transduction pathway as a target for cancer therapy. Oncogene. 2000 Dec 27;19(56):6680-6. doi: 10.1038/sj.onc.1204091. PMID 11426655
- [Background] Rowinsky EK. Targeting the molecular target of rapamycin (mTOR). Curr Opin Oncol. 2004 Nov;16(6):564-75. doi: 10.1097/01.cco.0000143964.74936.d1. PMID 15627018
- [Background] Blagosklonny MV, Darzynkiewicz Z. Four birds with one stone: RAPA as potential anticancer therapy. Cancer Biol Ther. 2002 Jul-Aug;1(4):359-61. No abstract available. PMID 12432246
- [Background] Gambacorti-Passerini CB, Gunby RH, Piazza R, Galietta A, Rostagno R, Scapozza L. Molecular mechanisms of resistance to imatinib in Philadelphia-chromosome-positive leukaemias. Lancet Oncol. 2003 Feb;4(2):75-85. doi: 10.1016/s1470-2045(03)00979-3. PMID 12573349
- [Background] Perry RA, Chamley JH, Robinson PM. Histochemically detected differences in cultured sympathetic neurons. J Anat. 1975 Jul;119(Pt 3):505-15. PMID 1141051
- [Background] Yu K, Toral-Barza L, Discafani C, Zhang WG, Skotnicki J, Frost P, Gibbons JJ. mTOR, a novel target in breast cancer: the effect of CCI-779, an mTOR inhibitor, in preclinical models of breast cancer. Endocr Relat Cancer. 2001 Sep;8(3):249-58. doi: 10.1677/erc.0.0080249. PMID 11566616
- [Background] Gibbons JJ, Discafani C, Peterson R, Hernandez R, Skotnicki J , Frost J. The Effect of CCI-779, a Novel Macrolide Antitumor Agent on the Growth of Human Tumor Cells in vitro and in Nude Mouse Xenograft in vitro. Proc. Am. Assoc. Cancer Res. 1999;40: Abstr. 2000.
- [Background] Geoerger B, Kerr K, Tang CB, Fung KM, Powell B, Sutton LN, Phillips PC, Janss AJ. Antitumor activity of the rapamycin analog CCI-779 in human primitive neuroectodermal tumor/medulloblastoma models as single agent and in combination chemotherapy. Cancer Res. 2001 Feb 15;61(4):1527-32. PMID 11245461
- [Background] Elit L. CCI-779 Wyeth. Curr Opin Investig Drugs. 2002 Aug;3(8):1249-53. PMID 12211424
- [Background] Teachey DT, Obzut DA, Cooperman J, Fang J, Carroll M, Choi JK, Houghton PJ, Brown VI, Grupp SA. The mTOR inhibitor CCI-779 induces apoptosis and inhibits growth in preclinical models of primary adult human ALL. Blood. 2006 Feb 1;107(3):1149-55. doi: 10.1182/blood-2005-05-1935. Epub 2005 Sep 29. PMID 16195324
- [Background] Peralba JM, DeGraffenried L, Friedrichs W, Fulcher L, Grunwald V, Weiss G, Hidalgo M. Pharmacodynamic Evaluation of CCI-779, an Inhibitor of mTOR, in Cancer Patients. Clin Cancer Res. 2003 Aug 1;9(8):2887-92. PMID 12912932
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu